CLINICAL TRIAL: NCT01091519
Title: Facts Study (Fakten-studie): Non-interventional Study to Investigate Whether Information Provided to Patients Influences Satisfaction With Toviaz Therapy As Perceived by the Patient
Brief Title: Non-Interventional Study To Investigate Whether Information Provided To Patients Influences Their Satisfaction With Toviaz Therapy
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221073; FACTS (FAKTEN) study
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: Non-interventional study fesoterodine educational materials
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Toviaz(fesoterodine) plus educational materials
  Interventions: Other: Toviaz(fesoterodine) plus educational materials
- Toviaz(fesoterodine) alone: Toviaz(fesoterodine) without additional educational materials
  Interventions: Other: Toviaz(fesoterodine) without educational materials

INTERVENTIONS:
Other: Toviaz(fesoterodine) plus educational materials — Educational materials including the Self-Assessment Goal Achievement (SAGA) tool to support dialogue.
  Groups: Toviaz(fesoterodine) plus educational materials
Other: Toviaz(fesoterodine) without educational materials — No educational materials
  Groups: Toviaz(fesoterodine) alone

SUMMARY:
Collect information on treatment with Toviaz (fesoterodine) under ordinary prescribing conditions, and to investigate whether additional educational information affects satisfaction with treatment as perceived by the patient.

DETAILED DESCRIPTION:
Patients will be identified and monitored during routine clinical practice visits, and will not be specifically selected as this would interfere with the representativeness of the results. The study will be conducted with office-based urologists and office-based general physicians, practitioners and internists (GPs) in Germany, thus representing a wide range of practices and populations. Each urologist or GP may invite patients to participate who have already been diagnosed with overactive bladder and prescribed Toviaz according to their usual standard of care. Study enrollment stopped on December 31, 2011 due to difficulty in recruiting patients. No safety issues were related to the decision to stop patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

Patients with increased urinary frequency and/or imperative urgency and/or urge incontinence, as can occur in patients with overactive bladder syndrome, for whom Toviaz was prescribed for treatment of the symptoms.

Patients will complete the OABv8 questionnaire and will need to meet a minimum score in order to be eligible for the study.

Exclusion Criteria:

Patients who meet the contraindications in the Toviaz prescribing information (active ingredient fesoterodine) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with overactive bladder symptoms presenting during routine clinical practice visits
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Schneider T, Arumi D, Crook TJ, Sun F, Michel MC. An observational study of patient satisfaction with fesoterodine in the treatment of overactive bladder: effects of additional educational material. Int J Clin Pract. 2014 Sep;68(9):1074-80. doi: 10.1111/ijcp.12450. Epub 2014 May 5. PMID 24797765
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221073&StudyName=Non-Interventional%20Study%20To%20Investigate%20Whether%20Information%20Provided%20To%20Patients%20Influences%20Their%20Satisfaction%20With%20Toviaz%20Therapy

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine With Educational Materials: Participants received prescription fesoterodine (Toviaz), which was guided by medical and therapeutic needs. Additionally all participants were provided with patient reported outcomes (PROs) for completion, with educational materials comprising of Self Assessment Goal Achievement (SAGA) tool. This tool included information to help the participants and follow their own treatment goals, as well as educational material on overactive bladder (OAB). Participants were observed for 4 months.
- Fesoterodine Without Educational Materials: Participants received prescription fesoterodine (Toviaz), which was guided by medical and therapeutic needs. Additionally all participants were provided with patient reported outcomes (PROs) for completion, without educational materials. Participants were observed for 4 months.
Period: Overall Study
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Started | 346 | 435
Treated | 342 | 431
Completed | 291 | 362
Not Completed | 55 | 73
Not completed — Adverse Event | 12 | 16
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 16 | 19
Not completed — Lost to Follow-up | 14 | 24
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 6 | 8
Not completed — Randomized not treated | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials | Total
Number analyzed (Participants) | 330 | 421 | 751
Age, Customized [Number; unit: participants] — For baseline characteristic age and gender, number of participants evaluable was 751.
  participants
    Less than (<) 18 years | 0 | 0 | 0
    18 to 44 years | 20 | 19 | 39
    45 to 64 years | 114 | 132 | 246
    Greater than or equal to (>=) 65 years | 196 | 270 | 466
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 263 | 502
  Male | 91 | 158 | 249

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Satisfied With Treatment at Month 4
Description: Participant's response to treatment was based on treatment satisfaction questionnaires (TSQ). Participants answered: "overall, how satisfied are you with your OAB medication?" and were asked to rate this question on 5 point scale as 1=very satisfied, 2=somewhat satisfied, 3= neither dissatisfied nor satisfied, 4=somewhat dissatisfied and 5=very dissatisfied. Five categorical responses were grouped to satisfied (including "very satisfied" and "somewhat satisfied") and dissatisfied (including "very dissatisfied", "somewhat dissatisfied", and "neither dissatisfied nor satisfied").
Time Frame: Month 4
Population: Full Analysis Set (FAS) included all participants who had received at least 1 dose of study medication and had provided at least 1 efficacy endpoint at baseline and during the study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Number analyzed (Participants) | 279 | 355
percentage of participants | 79.6 [74.4 to 84.1] | 76.1 [71.3 to 80.4]

2. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Week 4 and Month 4
Description: PPBC: single-item, self-administered validated questionnaire. Rated on a 6-point scale: participant was asked: "Which of the following statements describes your bladder condition best at the moment?" 1=no problems at all; 2=some very minor problems; 3=some minor problems; 4=some moderate problems; 5=severe problems; 6=many severe problems. Change from baseline results categorized as deterioration (Positive change from baseline); no Change (scores change=0); minor Improvement (negative score change in magnitude of 1); major improvement (negative score change in magnitude of >=2).
Time Frame: Baseline, Week 4, Month 4
Population: FAS included all participants who had received at least 1 dose of study medication and had provided at least 1 efficacy endpoint at baseline and during the study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. n=number of participants evaluable for this measure at specified time point.
Measure: Number; unit: participants
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Number analyzed (Participants) | 266 | 368
participants
  Baseline: No problem at all (n=266, 368) | 1 | 0
  Baseline: Some very minor problems (n=266, 368) | 2 | 3
  Baseline: Some minor problems (n=266, 368) | 15 | 16
  Baseline: Some moderate problems (n=266, 368) | 75 | 122
  Baseline: Severe problems (n=266, 368) | 145 | 179
  Baseline: Many severe problems (n=266, 368) | 28 | 48
  Change at Week 4: Deterioration (n=266, 368) | 12 | 14
  Change at Week 4: No change (n=266, 368) | 57 | 93
  Change at Week 4: Minor improvement (n=266, 368) | 90 | 107
  Change at Week 4: Major improvement (n=266, 368) | 107 | 154
  Change at Month 4: Deterioration (n=252, 330) | 7 | 4
  Change at Month 4: No change (n=252, 330) | 32 | 43
  Change at Month 4: Minor improvement (n=252, 330) | 49 | 82
  Change at Month 4: Major improvement (n=252, 330) | 164 | 201

3. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Urgency Scale (PPUS) at Week 4 and Month 4
Description: PPUS: single-item, self-administered validated questionnaire. Rated on a 3-point scale: participant was asked: "Which of the following would typically describe your experience when you have a desire to urinate?" 1=usually not able to hold urine; 2=usually able to hold urine (without leaking) until I reach a toilet if I go to the toilet immediately; 3= usually able to finish what I am doing before going to the toilet (without leaking). Change from baseline results categorized as deterioration (Negative change); no change (Score change=0); improvement (Positive change).
Time Frame: Baseline, Week 4, Month 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Number analyzed (Participants) | 252 | 351
participants
  Baseline: Usually not able hold urine (n=252, 351) | 75 | 116
  Baseline: Usually able to hold urine (n=252, 351) | 157 | 186
  Baseline: Usually able to finish (n=252, 351) | 20 | 49
  Change at Week 4: Deterioration (n=252, 351) | 19 | 28
  Change at Week 4: No Change (n=252, 351) | 130 | 174
  Change at Week 4: Improvement (n=252, 351) | 103 | 149
  Change at Month 4: Deterioration (n=238, 311) | 29 | 32
  Change at Month 4: No Change (n=238, 311) | 85 | 109
  Change at Month 4: Improvement (n=238, 311) | 124 | 170

4. Secondary Outcome: Number of Participants With Change From Baseline in Treatment Satisfaction Question (TSQ) at Week 4 and Month 4
Description: Participant's response to the treatment was based on treatment satisfaction questionnaires (TSQ). TSQ was rated on a 5-point scale, participant was asked: "overall how satisfied are you with your over active bladder (OAB) medication?" 1=very satisfied, 2=somewhat satisfied, 3=neither dissatisfied nor satisfied, 4=somewhat dissatisfied, 5=very dissatisfied. Change from baseline results categorized as deterioration (Positive change from baseline);no change (scores change=0);minor improvement (negative score change in magnitude of 1);major improvement (negative score change in magnitude of >=2).
Time Frame: Baseline, Week 4, Month 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Number analyzed (Participants) | 144 | 203
participants
  Baseline: Very Satisfied (n=144, 203) | 2 | 4
  Baseline: Somewhat Satisfied (n=144, 203) | 20 | 29
  Baseline:Neither Dissatisfied/Satisfied(n=144,203) | 47 | 54
  Baseline: Somewhat Dissatisfied (n=144, 203) | 60 | 95
  Baseline: Very Dissatisfied (n=144, 203) | 15 | 21
  Change at Week 4: Deterioration (n=144, 203) | 6 | 16
  Change at Week 4: No Change (n=144, 203) | 45 | 56
  Change at Week 4: Minor Improvement (n=144, 203) | 42 | 56
  Change at Week 4: Major Improvement (n=144, 203) | 51 | 75
  Change at Month 4: Deterioration (n=143, 179) | 2 | 10
  Change at Month 4: No Change (n=143, 179) | 33 | 38
  Change at Month 4: Minor Improvement (n=143, 179) | 51 | 48
  Change at Month 4: Major Improvement (n=143, 179) | 57 | 83

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE but distinct events are presented. An event may be categorized as serious in 1 subject, nonserious in another, or 1 subject may experience both serious, nonserious event. Safety population:participants who were randomized to with/without participant educational materials, had dose of prescription medication.
Arm/Group | Fesoterodine With Educational Materials | Fesoterodine Without Educational Materials
Serious Adverse Events (participants affected / at risk) | 2/342 | 1/431
Other Adverse Events (participants affected / at risk) | 25/342 | 36/431
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine With Educational Materials (N=342) | Fesoterodine Without Educational Materials (N=431)
Convulsion (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine With Educational Materials (N=342) | Fesoterodine Without Educational Materials (N=431)
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Accommodation disorder (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Oscillopsia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 3
Dry mouth (Gastrointestinal disorders) | 13 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse event (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This was an open label observational study in Germany, which was stopped early due to low participant recruitment rates. The results should therefore be interpreted with caution due to the lower than planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.